CLINICAL TRIAL: NCT06229210
Title: An Open-label, Multicenter Trial to Assess the Safety and Tolerability of Lumateperone in the Treatment of Pediatric Patients With Schizophrenia, Bipolar Disorder or Autism Spectrum Disorder
Brief Title: Safety and Tolerability Trial of Lumateperone in Pediatric Patients With Schizophrenia, Bipolar Disorder or Autism Spectrum Disorder
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Intra-Cellular Therapies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITI-007-321
Record Dates: First submitted 2024-01-19; First posted 2024-01-29 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Schizophrenia; Bipolar Disorder; Autism Spectrum Disorder
Keywords: Pediatric
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder; Autism Spectrum Disorder | interventions — lumateperone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lumateperone (Experimental)
  Interventions: Drug: Lumateperone

INTERVENTIONS:
Drug: Lumateperone — Lumateperone 5 mg - 42 mg capsules or orally disintegrating tablets administered orally, once daily based on age and indication

SUMMARY:
This is a multicenter, global, 26-week, open-label study to assess the safety and tolerability of lumateperone in pediatric patients with schizophrenia, bipolar disorder or autism spectrum disorder.

DETAILED DESCRIPTION:
The study will enroll pediatric patients as follows:

De Novo Patients:

* Patients with schizophrenia, including patients who have previously participated in the lumateperone open-label pediatric pharmacokinetic (PK) study (Study ITI-007-020)
* Patients with bipolar disorder who have previously participated in the lumateperone open-label pediatric PK study (Study ITI-007-030)
* Patients with irritability associated with autism spectrum disorder who have previously participated in the lumateperone open-label pediatric PK study (Study ITI-007-035)

Rollover Patients:

* Patients with bipolar disorder who are enrolling directly from a lead-in efficacy study.
* Patients with irritability associated with autism spectrum disorder who are enrolling directly from a lead-in efficacy study.

This study will be conducted as follows:

* A Screening Period of up to 2 weeks during which patient eligibility will be assessed.
* A 26-week Open-label Treatment Period (OLTP) during which all patients will receive open-label lumateperone once daily.
* A 2-week Safety Follow-up (SFU) Period: All patients should return to the clinic for the SFU visit approximately 2 weeks after the last dose of open-label lumateperone.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide consent as follows:

  * The patient's legally authorized representative (LAR) (eg, parent or guardian) must provide written, informed consent;
  * The patient must provide written assent to study enrollment;
* Male or female patients aged 13 to 17 years (inclusive) with schizophrenia; male or female patients aged 10 to 17 years (inclusive) with bipolar I or II disorder; or male or female patients aged 5 to 17 years (inclusive) with autism spectrum disorder;
* Meet Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition Text Revision (DSM-5-TR) primary diagnosis of schizophrenia, bipolar I or II disorder, or autism spectrum disorder as confirmed by Kiddie Schedule for Affective Disorders and Schizophrenia for School-Age Children-Present and Lifetime Version (K-SADS-PL).
* Is currently an outpatient and is anticipated to maintain outpatient status for the duration of the study.

Rollover Patients entering from the lead-in study must have safely completed the lead-in study, in the opinion of the Investigator.

Exclusion Criteria:

* Has a primary psychiatric diagnosis other than schizophrenia, bipolar I or bipolar II disorder or autism spectrum disorder. Schizophrenia with catatonia, or bipolar disorder with psychotic features are not allowed. Exceptions include:

  * ADHD: If a subject is taking psychostimulant(s) for ADHD, they must have been on a stable treatment regimen of these medication(s) for 30 days prior to Screening. The treatment regimen should remain stable throughout the study. This must be confirmed by the Investigator and noted in the source records.
  * For ASD patients only, based on Investigator opinion and DSM-5 criteria, mild or moderate intellectual disability is allowed. Severe or profound intellectual disability is exclusionary.
* In the opinion of the Investigator, the patient has a significant risk for suicidal behavior during their participation in the study or

  * At Screening, the patient scores "yes" on Suicidal Ideation Items 3, 4, or 5 of the Columbia-Suicide Severity Rating Scale (C SSRS) within 6 months prior to Screening or, at Baseline, the patient scores "yes" on Suicidal Ideation Items 3, 4, or 5 since the Screening Visit;
  * At Screening, the patient has had 1 or more suicidal attempts within the 2 years prior to Screening; or
  * At Screening or Baseline, scores > 3 on Item 13 (suicidal ideation) of the CDRS-R (for bipolar disorder patients only); or
  * The patient is considered to be an imminent danger to him/herself or others.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 500 (Estimated)
Dates: Start 2024-01-25 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Common Adverse Events | Up to 6 months
  An AE is any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug-related. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.

CONTACTS AND LOCATIONS:
Locations (43):
- United States (40):
  - Clinical Site, Phoenix, Arizona
  - Clinical Site, Little Rock, Arkansas
  - Clinical Site, Anaheim, California
  - Clinical Site, Colton, California
  - Clinical Site, Garden Grove, California
  - Clinical Site, Long Beach, California
  - Clinical Site, Redlands, California
  - Clinical Site, San Diego, California
  - Clinical Site, West Covina, California
  - Clinical Site, Colorado Springs, Colorado
  - Clinical Site, Gainesville, Florida
  - Clinical Site, Hialeah, Florida
  - Clinical Site, Miami, Florida
  - Clinical Site, Miami Gardens, Florida
  - Clinical Site, Miami Lakes, Florida
  - Clinical Site, Miami Springs, Florida
  - Clinical Site, Orlando, Florida
  - Clinical Site, Pompano Beach, Florida
  - Clinical Site, West Palm Beach, Florida
  - Clinical Site, Atlanta, Georgia
  - Clinical Site, Decatur, Georgia
  - Clinical Site, Lawrenceville, Georgia
  - Clinical Site, Savannah, Georgia
  - Clinical Site, Naperville, Illinois
  - Clinical Site, Indianapolis, Indiana
  - Clinical Site, Bloomfield Hills, Michigan
  - Clinical Site, Saint Charles, Missouri
  - Clinical Site, Lincoln, Nebraska
  - Clinical Site, Las Vegas, Nevada
  - Clinical Site, Avon Lake, Ohio
  - Clinical Site, Cincinnati, Ohio
  - Clinical Site, Garfield, Ohio
  - Clinical Site, Oklahoma City, Oklahoma
  - Clinical Site, Fort Worth, Texas
  - Clinical Site, Houston, Texas
  - Clinical Site, Plano, Texas
  - Clinical Site, Richmond, Texas
  - Clinical Site, Richmond, Virginia
  - Clinical Site, Bellevue, Washington
  - Clinical Site, Everett, Washington
- Serbia (3):
  - Clinical Site, Belgrade
  - Clinical Site, Niš
  - Clinical Site, Novi Sad

IPD SHARING:
Plan to Share IPD: No